CLINICAL TRIAL: NCT05740397
Title: Mean Arterial Pressure (MAP) Trial: Study Protocol for a Multicenter, Randomized, Controlled Trial to Compare Three Different Strategies of Mean Arterial Pressure Management During Cardiopulmonary By-pass
Brief Title: Trial to Compare Different Strategies of Mean Arterial Pressure Management During Cardiopulmonary By-pass
Acronym: MAP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliera Universitaria Integrata Verona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: "MAP" PROG.3048CESC
Record Dates: First submitted 2023-02-03; First posted 2023-02-23 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Heart; Surgery, Heart, Functional Disturbance as Result
Keywords: Cardiopulmonary by-pass

STUDY DESIGN:
Intervention Model Description: The present study is a randomized controlled three parallel groups trial. The patient allocation is 1:1:1. The outcome of patients undergoing cardiac surgery and treated with a MAP standard during CPB is compared to patients treated with high MAP and patient-tailored MAP during CPB
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard MAP (Other): Control group: MAP values between 50-60 mmHg
  Interventions: Other: Management of mean arterial pressure during cardiopulmonary by-pass in cardiac surgery interventions. The MAP will be mantained in the range of values of each study arm
- High MAP (Other): First Comparator group: MAP values between 70-80 mmHg
  Interventions: Other: Management of mean arterial pressure during cardiopulmonary by-pass in cardiac surgery interventions. The MAP will be mantained in the range of values of each study arm
- Patient-tailored MAP (Other): Second Comparator group: MAP comparable to the patient's pre-operative MAP. This one will be calculated by performing 3 blood pressure measurement in three different moments of the day before surgery (at 8 am, at 3 pm, and at 9 pm), and will be calculated using the standard formula "Diastolic AP + 0,33 x (systolic AP - Diastolic AP)". The preoperative MAP value obtained will be target during CPB, within a range of ± 10 mmHg
  Interventions: Other: Management of mean arterial pressure during cardiopulmonary by-pass in cardiac surgery interventions. The MAP will be mantained in the range of values of each study arm

INTERVENTIONS:
Other: Management of mean arterial pressure during cardiopulmonary by-pass in cardiac surgery interventions. The MAP will be mantained in the range of values of each study arm — The patients enrolled to elective cardiac surgeries will be evaluated during a pre-operative outpatient visit and widely informed about the chance to participate in the study. When patients undergo to the elective surgery general anaesthesia is administered and CPB is installed. The nominal flow for each patient will be 2,4 l/min/m2.
  To keep the MAP values around those corresponding to the randomized group, vasodilator (if MAP overcomes the assigned MAP value) or vasoconstrictor drugs will be used (if MAP value is lower than the assigned group). The following drugs will be used: nitroglicerine at incremental dose of 0,01 mcg/kg/min for a vasodilator effect and norepinephrine at incremental dose of 0,01 mcg/kg/min for a vasoconstrictor effect

SUMMARY:
* Background: One of the main goals of the Cardiopulmonary By-Pass (CPB) is targeting an adequate Mean Arterial Pressure (MAP), in order to maintain appropriate perfusion pressures in all end-organs during heart surgery. As inheritance of early studies, a value of 50-60 mmHg has been historically accepted as the "gold standard" MAP. However, in the last decades, the CPB management has remarkably changed, thanks to the evolution of technology and the availability of new biomaterials. Therefore, as already highlighted by the latest European Guidelines, the current management of CPB can no longer refer to those pioneering studies. To date, only few single-centre studies have compared different strategies of MAP management during CPB, but with contradictory findings and without achieving a real consensus. Therefore, what should be the ideal strategy of MAP management during CPB is still on debate. This trial will be the first multicentre, randomized, controlled study to compare three different strategies of MAP management during the CPB.
* Methods: We described herein the methodology of a multicenter, randomized, controlled trial comparing three different approaches to MAP targeting during CPB in patients undergoing elective cardiac surgery: the historically accepted "standard MAP" (50-60 mmHg), the "high MAP" (70-80 mmHg) and the "patient-tailored MAP" (comparable to the patient's preoperative MAP). It is the aim of the study to find the most suitable management in order to obtain the most adequate perfusion of end-organs during cardiac surgery. For this purpose, the primary endpoint will be the peak of serum lactate (Lmax) released during CPB, as index of tissue hypoxia. The secondary outcomes will include all the intraoperative parameters of tissues oxygenation and major post-operative complications related to organ malperfusion.
* Discussion: This trial will assess the best strategy to target the MAP during CPB to further improve the outcomes of cardiac surgery.

DETAILED DESCRIPTION:
Background:Most of cardiac surgery operations require a bloodless operating field and a steady heart (i.e. cardioplegic arrest). To ensure the perfusion of peripheral organs during the cardioplegic arrest time, the Cardipulmonary bypass (CPB) is installed. The CPB is a biomedical device, also named Heart-Lung machine, that, through a circuit, filtrates and oxygenates venous blood coming from the patient, giving it back as arterial blood through a mechanical pump. The blood flow produced by the CPB is continuous, then the pressure produced is a Mean Arterial Pressure (MAP). The MAP can be modulated by vasoactive and/or anaesthetic drugs during CPB, in order to maintain an appropriate perfusion pressures in all end-organs, avoiding tissue hypoperfusion and hypoxia. The latter, indeed, may occur in the post-operative period as organ damage: cerebral ischemia and consequently transitory or permanent neurological injury, renal ischemia and consequently acute kidney injury, or gastrointestinal ischemia. Consequently, the management of MAP acquires a crucial role. A value of 50-60 mmHg has been historically accepted as the "gold standard" MAP, according to the early experiments and pioneering cardiac surgery investigations. However, in the last decades, the CPB has remarkably changed thanks to the evolution of technology and availability of new biomaterials. Therefore, as already highlighted by the latest European Guidelines, the current management of CPB can no longer refer to those pioneering studies. To date, only few single-center studies focused their attention on the correlation between MAP values during CPB and cardiac surgery outcomes. One study compared the "high-target" MAP (70-80 mmHg) to "standard" MAP (50-60 mmHg) in terms of new post-operative cerebral injuries. They reported a higher incidence of stroke (7.0% vs 1.1%; P=0.09) and mortality (4.1% vs 0%; P=0.06) in the "high-target" MAP population compared to the "low-target" group. Conversely, another author, reported a reduction (from 12.9% to 4.8%) of major cardiac and neurologic events in patients treated with higher MAP compared to patients treated with the "standard" MAP during coronary artery bypass graft surgery (CABG). However, they are both single-center studies, with small sample sizes; moreover, the second one involves only CABG patients. Finally, a third author compared the "high-MAP" (80 mmHg) with "patient-tailored" MAP (comparable to pre-operative MAP in the single patient). The study showed no differences in terms of major cardiac and neurologic events (11.7% and 12.6% respectively), but also the study included only patients undergoing CABG surgery. However, all the above-mentioned studies showed conflicting evidences, without achieving a real consensus on what should be the most adequate MAP target during CPB.

The purpose of our randomized study is to define the best strategy to obtain an "ideal MAP" during CPB, comparing the historically accepted "standard MAP" (50-60 mmHg) with the "high MAP" (70-80 mmHg) and with the "patient-tailored MAP". To investigate the risk of hypoperfusion and to evaluate whether the MAP during CPB is adequate to avoid tissue hypoxia, the serum lactate value will be collected at different time-points, as index of tissue anaerobiosis/hypoperfusion. To date, several studies have analysed the trend of lactates intraoperatively and postoperatively, and hyperlactatemia demonstrated to be a predictive factor of post-operative mortality and morbidity. Particularly, some authors describe that a peak of lactates > 4 mmol/l during CPB relates to post-operative mortality. Another study considered a cut-off of 3 mmol/l, and also in this case, hyperlactatemia during CPB relates to post-operative major complications. However, both studies do not give information about the precise value of lactates reached, neither about the entire trend of lactates released during CBP. Therefore, differently from previous studies, the primary endpoint of this trial will be the peak value (absolute value) of serum lactates (Lmax) measured during CPB.

Methods: Participants, interventions and outcomes Study setting:Coordinator centre: Division of Cardiac Surgery, Azienda Ospedaliera Universitaria Integrata Verona, Italy.

Participating Centers:Center 1: Division of Cardiac Surgery at Ospedale Maggiore, Parma, Italy; Center 2: Division of Cardiac Surgery at Azienda Sanitaria Universitaria Friuli Centrale, Udine, Itay.Center 3: Division of Cardiac Surgery at Hospital Clinic de Barcelona, Barcelona, Spain Intervention description:The treatment groups will be:Group 1: Standard MAP: MAP values between 50-60 mmHg as control group. Group 2: High MAP: MAP values between 70-80 mmHg. Group 3: Patient-tailored MAP: MAP comparable to the patient's pre-operative MAP.

Procedures,Preoperative: Day before surgery:

* Collection of informed consent for participating the study
* Randomization
* Measurement of preoperative MAP in every patient enrolled, regardless of the assignment group through randomization.
* Blood samples to assess: Hemoglobin , Hematocrit, white blood cells , platelets , C reactive protein, lactate dehydrogenase , prothrombin time , activated partial thromboplastin time, fibrinogen and creatinine, lipase, pancreatic amylase, alanina aminotransferase, aspartate aminotransferase, total bilirubin, conjugated bilirubin, unconjugated bilirubin, gamma-glutamyltransferase, alkaline phosphatase ) and albumin
* Arterial blood gas test to evaluate preoperative lactatemia
* Calculation of eGFR (according to MDRD) to evaluate preoperative renal function
* Evaluation of preoperative mRS in case of stroke in amnestic history. Intraoperative
* Intraoperative monitoring of MAP during CPB: at the beginning of CPB, every 20 minutes until minute 300 and at the end of CPB.
* ABG after orotracheal intubation, at the beginning of CPB, every 20 minutes during ECC (eventually until minute 300), at the end of CPB, at the end of surgery. Data collected: lactates as organ perfusion index, Hb and Hct.
* Real time and continuous monitoring of respiratory gases during CPB suggestive of the perfusion trend, through CDI ® 550 Blood parameter monitoring system (Terumo Europe), data collection related to Oxygen Delivery, Oxygen consumption e Oxygen extraction, at the beginning of CPB, every 20 minutes (until minute 300) and at the end of CPB.
* Intraoperative monitoring of Near-Infrared Spectroscopy, NIRS defined as non-invasive measurement of cerebral microcirculatory blood flow. Data will be collected at anesthesia induction, before skin incision, at the beginning of CPB, every 20 minutes (until minute 300), at the end of CPB and at the end of surgery.
* Monitoring of CPB and aortic cross-clamp times
* Calculation of "Vasoactive-inotropic score" (VIS) which relates the entity of inotropic and or vasoactive support.

Postoperative:

Post-operavtive day (POD) at arrival in Intensive Care Unit (ICU), POD 1 and 4:

* Blood chemistry samples
* Calculation of eGFR (according to MDRD)
* ABG at arrival in ICU, at 3-6-12-24 hours after surgery. Data collection on: serum lactates, pH, paO2, paCO2, BE, HCO3-, calculation of the Pa/Fi ratio
* Chest X-ray and evaluation of eventual pulmonary damage through Murray "Lung Injury Score" (LIS)
* Monitoring of extubation time (hours)
* Calculation of VISmax
* Monitoring of postoperative cardiac function at POD 4 through the evaluation of LVEF
* Monitoring of postoperative stroke through the "modified Rankin Scale" (mRS).
* Evaluation of acute kidney injury through the definition of "Acute Kidney Injury" (AKIN)
* Monitoring of gastrointestinal ischemia
* Monitoring of in-hospital death

Follow-up visit at 30 days from surgery:

* mRS score
* eGFR and AKIN score
* LVEF
* Re-hospitalization
* Death for cardiovascular or other causes. All the procedures listed above are considered the standard of care in the clinical practice at the Cardiac Surgery Divisions of all the Participating Centres.

If any of the following clinical situations occur during the study period in patients already enrolled, this will be reason for exclusion of the patient from the study: withdrawal of consent by the patient, unplanned additional procedures, necessary during surgery for complications in itinere (not provided in the preoperative planning), the need of mechanical circulatory support > 72 hours.

Sample size:The sample size has been calculated for the primary endpoint: the maximum serum lactate value (Lmax). A preliminary analysis was performed on a sample size of 128 consecutive patients undergone to elective cardiac surgery at Cardiac Surgery Division at AOUI of Verona (about the 10% of the annual volume cases at our Institution). All patients were treated with standard MAP (standard of care) and the estimated mean of Lmax during CPB was 1.25 mmol/l, with a standard deviation of 0.7 mmol/l. Starting from this value, a reduction of -15% of the mean Lmax was considered clinically significant for every comparison that will be performed in the study:Standard MAP vs High MAP (-15%) difference d=-0,19; Standard MAP vs patient-tailored MAP (-15%) difference d=-19;High MAP vs patient-tailored MAP (-15%) difference d=-19. Based on these assumptions, performing the Mann-Whitney non-parametric test and considering an alpha of 0.05 sec. Bonferroni for all the three comparisons (corrected Alpha= 0.01667) and a power of 80%, 300 patients should be enrolled for each group, for a total of 900 patients (PASS 14). To account for a potential drop-out of 10%, the size becomes 333 patients per group, then a total of 999 patients. The number of patients that each Participating Centres should recruit, has been calculated based on the annual cases volume of each Centre: AOUI Verona: 327 cases (109 per group); Ospedale Maggiore di Parma: 162 cases (54 per group); Azienda Sanitaria Universitaria Friuli Centrale di Udine: 231 cases (77 per group); Hospital Clinic de Barcelona, Spain: 279 cases (93 per group). Patients will be recruited at Cardiac Surgery Division of each Participating Centre. Recruitment will continue until the expected total number of patients will be reached. The list of randomization will be generated for each centre using STATA statistical software 14, by the Clinical Research Unit of Azienda Ospedaliera Universitaria Integrata of Verona. The balanced blocks randomization method will be used. The block size will be of 6,9 or 12 according to the number of treatment groups.

Data collection and management: All preoperative, intraoperative and post-operative procedures are standard of care in each Cardiac Surgery Division. The data collection will take place during the patient hospitalization by the research team in a dedicated datasheet. All the data are listed in the protocol and will be retrieved from the Hospital health information system. A separated datasheet with the same coding will be used for the Participating Centers. At the end of the study, all datasheets will be unified in a unique database and analysed by the Promoting Center. Research data will be stored using a study identification code for each participant. The key to the identification code list will only be available to the research team during the study and will be documented and safeguarded by the principal investigator according to research guidelines after completion of the study. No patient identification details will be reported in publications. Data collection and management will be in accordance with the EU regulation 2016/679, the Privacy Code (D.lgs 196/03 s.m.i ), and Guide Lines of 24th July 2008, and will be guaranteed by the promoter of the study. The Promoter will store the original paper documentations for at least 7 years in compliance with LD 200/2007.

Statistical methods:Demographic and clinical characteristics will be presented as percentage in case of ordinal variables and as percentages, means, medians and standard deviations and/or interquartile range in case of categorical and/or quantitative variables. The Pearson χ 2 and the H-test by Kruskall Wallis will be used for any assessment of differences between the three groups. To evaluate the primary endpoint of the study the Mann-Whitney test will be used for comparisons between groups with an alpha equal to 0.01667. The Mann-Whitney test will also be used to evaluate the secondary endpoint obtained by AUC, while the Pearson χ 2 will be used to compare the proportion of cases above and below the serum lactate peak cut-off > 3mmol. To compare the secondary endpoints in the three groups according to the types of variables, ANOVA or non-parametric H-test by Kruskall Wallis will be used for quantitative variables, while Pearson χ 2 test will be performed for dichotomous or categorical variables. ANOVA for repeated measures, or Friedman test or the mixed effects model will be used for variables collected at different timepoints. A p-value < 0.05 will be considered statistically significant . Both an Intention to treat (ITT) and per protocol (PP) analysis will be performed. Missing data will be handled by different data imputation methods (IPW-inverse probability weighting and LCOF-Last-Observation-Carried-Forward method) with sensitivity analysis.

Oversight and monitoring: The Promoter will have the responsibility for the study management. The data monitoring committee will be constituted by the Promoter and the Principal investigators of the Participating Centres who will meet twice a year to check the appropriateness of the investigation, by checking the data of a minimum of 40% of the patients. Any changes to the study protocol will be communicated to the AOUI of Verona Institutional Review Board and the Regional Ethical Committees responsible for approving the study.

ELIGIBILITY:
Inclusion Criteria:

* Elective surgery
* Index of surgical risk Euroscore II < 9%
* The following procedures will be considered: Isolated or combined with aortic or mitral valve surgery coronary artery bypass graft surgery for acute or chronic coronary artery disease isolated aortic valve replacement for aortic stenosis and/or aortic regurgitation ; isolated mitral valve repair or replacement for mitral stenosis and/or mitral regurgitation; isolated ascending aorta surgery with or without aortic valve replacement
* Surgical approach through complete and/or mini-sternotomy
* Preserved or mildly reduced left ventricular ejection fraction (LVEF ≥ 40%) at preoperative echocardiography
* Patients with an estimated Glomerular filtration rate (eGFR) ≥ 40 ml/min/mq calculated using the Modification of Diet in Renal Disease formula (MDRD)
* Signed informed consent

Exclusion Criteria:

* Age < 18 years and >80 years
* Reoperation
* Emergent, urgent and salvage procedures
* Euroscore II > 9%
* Right toracothomy procedures
* Any surgical procedure not listed above (i.e. tricuspid valve surgery, aortic root surgery, congenital heart diseases, surgery necessitating hypotermic circulation arrest, surgical ablation of atrial fibrillation etc.)
* More than mild left ventricular dysfunction at preoperative echocardiogram (LVEF < 40%)
* Patients with critical preoperative state: any ventricular fibrillation or ventricular tachycardia, preoperative cardiac massage, preoperative ventilation before anaesthetic room, preoperative inotropes or mechanical circulatory support planned before cardiac intervention (i.e. during coronary angiography) and other conditions according to Euroscore II definition.
* Patients with an estimated eGFR < 40 ml/min/mq calculated using the MDRD or patients on dialysis.
* Patients with chronic obstructive pulmonary disease > 3 stage according to Global Initiative for Chronic Obstructive Lung Disease (GOLD) 2019 classification.
* Patients with severe preoperative epatic failure (CHILD-PUGH ≥ B)
* Patient with severe symptomatic carotid atheromasia

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 900 (Estimated)
Dates: Start 2021-05-03 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Serum lactate peak (Lmax) (mmol/l) detected during Cardiopulmonary by-pass time | at the beginning of CPB, every 20 minutes during CPB, at the end of CPB, at the end of surgery
  The mean of this value will be compared in the three groups of treatment.

SECONDARY OUTCOMES:
The area under the curve (AUC) of the serum lactate values measured during CPB | at the beginning of CPB, every 20 minutes during CPB, at the end of CPB, at the end of surgery
  The area under the curve (AUC) of the serum lactate values measured during CPB
Number of cases with serum lactate peak > 3 mmol/l during CPB | at the beginning of CPB, every 20 minutes during CPB, at the end of CPB, at the end of surgery
  Number of cases with serum lactate peak > 3 mmol/l during CPB
Evaluation of intraoperative cerebral perfusion (through monitoring of NIRS) | at anesthesia induction, before skin incision, at the beginning of CPB, every 20 minutes (until minute 300), at the end of CPB and at the end of surgery.
  Near-Infrared Spectroscopy NIRS (23) defined as non-invasive measurement of cerebral microcirculatory blood flow
Intraoperative pulmonary perfusion (through Pa/Fi ratio, paO2, paCO2 at ABG and VO2R and DO2 of CDI) | at the beginning of CPB, every 20 minutes (until minute 300) and at the end of CPB.
  CDI ® 550 Blood parameter monitoring system (Terumo Europe) (22), data collection related to Oxygen Delivery (DO2), Oxygen consumption (VO2) e Oxygen extraction (O2ER), at the beginning of CPB, every 20 minutes (until minute 300) and at the end of CPB
Evaluation of intraoperative and postoperative low cardiac output syndrome (through the calculation of VISmax) | at the beginning of CPB, every 20 minutes (until minute 300) and at the end of CPB.
  Vasoactive-inotropic score" (VIS) (24) which relates the entity of inotropic and or vasoactive support. VIS max is obtained through the following calculation: [Dopamine dose (mcgkg/min)+ Dobutamine dose (mcg/kg/min) + 100 x Epinephrine dose (mcg/kg/min) + 50 x Levosimendan dose (mcg/kg/min) + 10 x Milrinone dose (mcg/kg/min) + 10,000 x Vasopressin dose (units/kg/min) + 100 x Norepinephrine dose (mcg/kg/min)]. The VIS will be calculated according to the length of surgery
Postoperative and 30-day LVEF (%) | at 1 hour from the end of the operation, at 12 hours and at 96 hours after the end of the operation
  Post-operative echocardiography
Evaluation of pulmonary injury (through the LIS) | at 1 hour from the end of the operation, at 12 hours and at 96 hours after the end of the operation
  "Lung Injury Score" (LIS) (25). The score considers 4 criteria for the development of ALI/ARDS: Hypoxemia, respiratory system compliance, chest radiographic findings and the positive expiratory pressure level. Each criteria receives a score from 0 to 4 according to the gravity of the condition. The final score is obtained dividing the collective score by the number of components used. A score equal to 0 shows the absence of pulmonary damage, a score between 1 and 2.5 shows a mild to moderate pulmonary damage and a final score major than 2.5 shows the presence of ARDS
Postoperative and 30-day Acute Kidney Injury (according to AKIN score) | at 1 hour from the end of the operation, at 12 hours and at 96 hours after the end of the operation
  Acute Kidney Injury" (AKIN) (27) through a stratification of renal damage in three stages: 1) Creatinine × 1.5 - 2.0 from baseline or Creatinine increased by at least 0,3 mg/dl (26.5μmol/L); 2) Creatinine × 2.0-2.9 from baseline; 3) Creatinine > 3.0 from baseline or Creatinine increased at least 4 mg/dl (353.6 umol/l) or the initiation of dialysis
Postoperative gastrointestinal ischemia | at 1 hour from the end of the operation, at 12 hours and at 96 hours after the end of the operation
  a diagnosed ischemia by a surgery consultant according to the value of serum lactate, WBC, clinical and radiological (CT scan and/or abdomen ultrasound) examination.
Hepatic function and coagulation indexes | at 1 hour from the end of the operation, at 12 hours and at 96 hours after the end of the operation
  prothrombin time (PT/INR), activated partial thromboplastin time (aPTT), fibrinogen and creatinine (mg/dl), lipase, pancreatic amylase, alanine aminotransferase (ALT), aspartate aminotransferase (AST), total bilirubin (Bil Tot), conjugated bilirubin (direct Bil), unconjugated bilirubin (indirect Bil), gamma-glutamyltransferase (GGT), alkaline phosphatase (ALP) and albumin
Evaluation of neurological dysfunction | at 1 hour from the end of the operation, at 12 hours and at 96 hours after the end of the operation
  (as dichotomous variable) and evaluation through mRS (0-6) in case permanent neurological injury
In-hospital mortality and at 30 days from surgery | At 30 days after the operation
  Death (dichotomous variable)

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliera Universitaria Integrata di Verona, Verona, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Puis L, Milojevic M, Boer C, De Somer FMJJ, Gudbjartsson T, van den Goor J, Jones TJ, Lomivorotov V, Merkle F, Ranucci M, Kunst G, Wahba A; EACTS/EACTA/EBCP Committee Reviewers. 2019 EACTS/EACTA/EBCP guidelines on cardiopulmonary bypass in adult cardiac surgery. Interact Cardiovasc Thorac Surg. 2020 Feb 1;30(2):161-202. doi: 10.1093/icvts/ivz251. No abstract available. PMID 31576402
- [Background] Hecker BR, Knopes KD. Optimal pressures and flows during cardiopulmonary bypass. Con: pressure is more important than flow. J Cardiothorac Vasc Anesth. 1991 Aug;5(4):402-4. doi: 10.1016/1053-0770(91)90169-t. No abstract available. PMID 1873521
- [Background] Evans RG, Lankadeva YR, Cochrane AD, Marino B, Iguchi N, Zhu MZL, Hood SG, Smith JA, Bellomo R, Gardiner BS, Lee CJ, Smith DW, May CN. Renal haemodynamics and oxygenation during and after cardiac surgery and cardiopulmonary bypass. Acta Physiol (Oxf). 2018 Mar;222(3). doi: 10.1111/apha.12995. Epub 2017 Nov 30. PMID 29127739
- [Background] Andersson LG, Bratteby LE, Ekroth R, Hallhagen S, Joachimsson PO, van der Linden J, Wesslen O. Renal function during cardiopulmonary bypass: influence of pump flow and systemic blood pressure. Eur J Cardiothorac Surg. 1994;8(11):597-602. doi: 10.1016/1010-7940(94)90043-4. PMID 7893500
- [Background] Byhahn C, Strouhal U, Martens S, Mierdl S, Kessler P, Westphal K. Incidence of gastrointestinal complications in cardiopulmonary bypass patients. World J Surg. 2001 Sep;25(9):1140-4. doi: 10.1007/BF03215861. PMID 11571949
- [Background] Nilsson J, Hansson E, Andersson B. Intestinal ischemia after cardiac surgery: analysis of a large registry. J Cardiothorac Surg. 2013 Jun 18;8:156. doi: 10.1186/1749-8090-8-156. PMID 23777600
- [Background] Murphy GS, Hessel EA 2nd, Groom RC. Optimal perfusion during cardiopulmonary bypass: an evidence-based approach. Anesth Analg. 2009 May;108(5):1394-417. doi: 10.1213/ane.0b013e3181875e2e. PMID 19372313
- [Background] GLIEDMAN ML, LEWIS FJ, SHUMWAY NE. A mechanical pump-oxygenator for successful cardiopulmonary by-pass. Surgery. 1956 Nov;40(5):831-9. No abstract available. PMID 13371445
- [Background] ABRAMS LD. The practice of total cardio-pulmonary by-pass; a short review. Postgrad Med J. 1959 Mar;35(401):144-6 passim. doi: 10.1136/pgmj.35.401.144. No abstract available. PMID 13633628
- [Background] SCURR CF. Cardio-pulmonary by-pass: physiological considerations. Proc R Soc Med. 1958 Aug;51(8):581-9. No abstract available. PMID 13578951
- [Background] Slogoff S, Reul GJ, Keats AS, Curry GR, Crum ME, Elmquist BA, Giesecke NM, Jistel JR, Rogers LK, Soderberg JD, et al. Role of perfusion pressure and flow in major organ dysfunction after cardiopulmonary bypass. Ann Thorac Surg. 1990 Dec;50(6):911-8. doi: 10.1016/0003-4975(90)91118-u. PMID 2241382
- [Background] Vedel AG, Holmgaard F, Rasmussen LS, Langkilde A, Paulson OB, Lange T, Thomsen C, Olsen PS, Ravn HB, Nilsson JC. High-Target Versus Low-Target Blood Pressure Management During Cardiopulmonary Bypass to Prevent Cerebral Injury in Cardiac Surgery Patients: A Randomized Controlled Trial. Circulation. 2018 Apr 24;137(17):1770-1780. doi: 10.1161/CIRCULATIONAHA.117.030308. Epub 2018 Jan 16. PMID 29339351
- [Background] Gold JP, Charlson ME, Williams-Russo P, Szatrowski TP, Peterson JC, Pirraglia PA, Hartman GS, Yao FS, Hollenberg JP, Barbut D, et al. Improvement of outcomes after coronary artery bypass. A randomized trial comparing intraoperative high versus low mean arterial pressure. J Thorac Cardiovasc Surg. 1995 Nov;110(5):1302-11; discussion 1311-4. doi: 10.1016/S0022-5223(95)70053-6. PMID 7475182
- [Background] Charlson ME, Peterson JC, Krieger KH, Hartman GS, Hollenberg JP, Briggs WM, Segal AZ, Parikh M, Thomas SJ, Donahue RG, Purcell MH, Pirraglia PA, Isom OW. Improvement of outcomes after coronary artery bypass II: a randomized trial comparing intraoperative high versus customized mean arterial pressure. J Card Surg. 2007 Nov-Dec;22(6):465-72. doi: 10.1111/j.1540-8191.2007.00471.x. PMID 18039205
- [Background] Weil MH, Afifi AA. Experimental and clinical studies on lactate and pyruvate as indicators of the severity of acute circulatory failure (shock). Circulation. 1970 Jun;41(6):989-1001. doi: 10.1161/01.cir.41.6.989. No abstract available. PMID 5482913
- [Background] Boldt J, Piper S, Murray P, Lehmann A. Case 2-1999. Severe lactic acidosis after cardiac surgery: sign of perfusion deficits? J Cardiothorac Vasc Anesth. 1999 Apr;13(2):220-4. doi: 10.1016/s1053-0770(99)90093-9. No abstract available. PMID 10230962
- [Background] TRANQUADA RE. LACTIC ACIDOSIS. Calif Med. 1964 Dec;101(6):450-61. No abstract available. PMID 14232165
- [Background] OLSON RE. "EXCESS LACTATE" AND ANAEROBIOSIS. Ann Intern Med. 1963 Dec;59:960-3. doi: 10.7326/0003-4819-59-6-960. No abstract available. PMID 14082746
- [Background] Minton J, Sidebotham DA. Hyperlactatemia and Cardiac Surgery. J Extra Corpor Technol. 2017 Mar;49(1):7-15. PMID 28298660
- [Background] Demers P, Elkouri S, Martineau R, Couturier A, Cartier R. Outcome with high blood lactate levels during cardiopulmonary bypass in adult cardiac operation. Ann Thorac Surg. 2000 Dec;70(6):2082-6. doi: 10.1016/s0003-4975(00)02160-3. PMID 11156124
- [Background] Ranucci M, De Toffol B, Isgro G, Romitti F, Conti D, Vicentini M. Hyperlactatemia during cardiopulmonary bypass: determinants and impact on postoperative outcome. Crit Care. 2006;10(6):R167. doi: 10.1186/cc5113. PMID 17134504
- [Background] Newland RF, Baker RA, Stanley R. Electronic data processing: the pathway to automated quality control of cardiopulmonary bypass. J Extra Corpor Technol. 2006 Jun;38(2):139-43. PMID 16921687
- [Background] Brady K, Joshi B, Zweifel C, Smielewski P, Czosnyka M, Easley RB, Hogue CW Jr. Real-time continuous monitoring of cerebral blood flow autoregulation using near-infrared spectroscopy in patients undergoing cardiopulmonary bypass. Stroke. 2010 Sep;41(9):1951-6. doi: 10.1161/STROKEAHA.109.575159. Epub 2010 Jul 22. PMID 20651274
- [Background] Yamazaki Y, Oba K, Matsui Y, Morimoto Y. Vasoactive-inotropic score as a predictor of morbidity and mortality in adults after cardiac surgery with cardiopulmonary bypass. J Anesth. 2018 Apr;32(2):167-173. doi: 10.1007/s00540-018-2447-2. Epub 2018 Jan 13. PMID 29332153
- [Background] Asimakopoulos G, Smith PL, Ratnatunga CP, Taylor KM. Lung injury and acute respiratory distress syndrome after cardiopulmonary bypass. Ann Thorac Surg. 1999 Sep;68(3):1107-15. doi: 10.1016/s0003-4975(99)00781-x. PMID 10510030
- [Background] Banks JL, Marotta CA. Outcomes validity and reliability of the modified Rankin scale: implications for stroke clinical trials: a literature review and synthesis. Stroke. 2007 Mar;38(3):1091-6. doi: 10.1161/01.STR.0000258355.23810.c6. Epub 2007 Feb 1. PMID 17272767
- [Background] Khwaja A. KDIGO clinical practice guidelines for acute kidney injury. Nephron Clin Pract. 2012;120(4):c179-84. doi: 10.1159/000339789. Epub 2012 Aug 7. No abstract available. PMID 22890468
- [Derived] Francica A, Mazzeo G, Galeone A, Linardi D, San Biagio L, Luciani GB, Onorati F. Mean Arterial Pressure (MAP) Trial: study protocol for a multicentre, randomized, controlled trial to compare three different strategies of mean arterial pressure management during cardiopulmonary bypass. Trials. 2024 Mar 15;25(1):191. doi: 10.1186/s13063-024-07992-3. PMID 38491507